CLINICAL TRIAL: NCT06311955
Title: Prospective Phase II Clinical Study of Postoperative Carbon Ion Radiotherapy for Thymic Epithelial Malignant Tumor Received R2 Resection
Brief Title: Clinical Study of Postoperative Carbon Ion Radiotherapy for Thymus Tumor With Residual Tumor
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jian Chen (Other)
Responsible Party: Sponsor-Investigator, Jian Chen, Clinical Professor, Shanghai Proton and Heavy Ion Center
Organization: Shanghai Proton and Heavy Ion Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPHIC-TR-THLC2023-06
Record Dates: First submitted 2024-03-09; First posted 2024-03-15 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Thymic Epithelial Tumor; Radiotherapy Side Effect; Carbon Ion Radiotheray; Heavy Ion Radiotherapy
MeSH Terms: conditions — Thymic epithelial tumor; Radiation Injuries | interventions — Heavy Ion Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study arm (Experimental): The patients will receive 72GyE per 18 fractions of carbon ion radiotherapy. Patients with thymus cancer should be combined with platinum-based regimen (including etoposide combined with cisplatin / carboplatin / loplatin / nedaplatin; paclitaxel combined with cisplatin or cisplatin / carboplatin / loplatin / nedaplatin; docetaxel combined with cisplatin / carboplatin / loplatin / nedaplatin) for at least 4 cycles. The primary endpoint was progression-free survival and toxicities, and the secondary endpoint was local relapse-free survival, overall survival and cause-specific survival.
  Interventions: Radiation: Carbon ion radiotherapy; Other: combined with platinum-based regimen

INTERVENTIONS:
Radiation: Carbon ion radiotherapy — The patients will receive 72GyE per 18 fractions of carbon ion radiotherapy. Patients with thymus cancer should be combined with platinum-based regimen (including etoposide combined with cisplatin / carboplatin / loplatin / nedaplatin; paclitaxel combined with cisplatin or cisplatin / carboplatin / loplatin / nedaplatin; docetaxel combined with cisplatin / carboplatin / loplatin / nedaplatin) for at least 4 cycles. The primary endpoint was progression-free survival and toxicities, and the secondary endpoint was local relapse-free survival, overall survival and cause-specific survival.
Other: combined with platinum-based regimen — combined with platinum-based regimen

SUMMARY:
To observe the efficacy and toxicities of heavy ion radiation therapy for locally advanced or advanced primary thymic epithelial malignant tumor received R2 resection. The primary endpoint was progression-free survival and toxicities, and the secondary endpoint was local relapse-free survival, overall survival and cause-specific survival.

DETAILED DESCRIPTION:
The patients will receive 72GyE per 18 fractions of carbon ion radiotherapy. Patients with thymus cancer should be combined with platinum-based regimen (including etoposide combined with cisplatin / carboplatin / loplatin / nedaplatin; paclitaxel combined with cisplatin or cisplatin / carboplatin / loplatin / nedaplatin; docetaxel combined with cisplatin / carboplatin / loplatin / nedaplatin) for at least 4 cycles. The primary endpoint was progression-free survival and toxicities, and the secondary endpoint was local relapse-free survival, overall survival and cause-specific survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage II-IV (Masaoka-Koga) thymus epithelial malignancies without a history of thoracic radiotherapy who had undergone radical surgery (R2 resection, visible residual tumor) and had a definite pathological diagnosis.
* Sign informed consent.
* Between the ages of 18 and 70.
* ECOG general status score of 0-2.
* The expected survival is at least 6 months.
* Adequate organ function: 1). Blood function: absolute neutrophil count (ANC) ≥1.5 x 109/L, platelet count ≥80 x 109/L, hemoglobin ≥9 g/dL 2). Lung function: FEV1>25%, DLCO>25% 3). Cardiac function: no serious pulmonary hypertension, cardiovascular and cerebrovascular diseases, peripheral vascular diseases, serious chronic heart disease and other complications that may affect radiotherapy.4). Adequate liver function: total bilirubin <1.5 times the upper limit of normal value, and AST, ALT<2 times the upper limit of normal value. 5). Adequate renal function: serum creatinine ≤1.5 times the upper limit of normal or calculated creatinine clearance ≥50 ml /min, and urinary protein <2+. Patients with a baseline urinary protein level of 2+ or more should have a 24-hour urine collection and evidence of a 24-hour urinary protein level of 1g or less.

Exclusion Criteria:

* Complicated with other malignant tumors that have not been controlled.
* Have large quantity of pleural or pericardial effusion.
* Patient whose particle radiotherapy plan cannot meet the minimum target dose coverage and dose volume limitation requirements, or cannot meet the dose constrains of normal tissue or organs.
* Chest radiation therapy or radioactive particle implantation history.
* Cardiac pacemakers or other internal metal prosthesis implants that may be affected by high-energy radiation or may affect the dose distribution to the radiation target area.
* Pregnancy (confirmed by serum or urine β-HCG test) or lactation period.
* HIV positive. Hepatitis virus replication phase, need to receive antiviral therapy, but because of concomitant disease cannot receive antiviral therapy. Active stage of syphilis.
* A history of mental illness may hinder the completion of treatment.
* With serious comorbidity that may interfere with radiotherapy, including: (a) Acute infectious diseases or acute active phase of chronic infection. b) Unstable angina pectoris, congestive heart failure, myocardial infarction that has been hospitalized in the past 6 months. c) Exacerbations of chronic obstructive pulmonary disease or other respiratory conditions requiring hospitalization. d) Severely impaired immune function. e) Diseases with excessive sensitivity to radiation such as ataxia telangiectasia. f) Other diseases that may affect particle radiotherapy.
* Other circumstances that the physician considers inappropriate to participate in clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Disease progression-free survival rate | From date of radiotherapy started until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  Disease progression-free survival rate was defined from the start of carbon ion radiotherapy till the date of disease progression at any site or death, or the last follow up.
Incidence of Treatment-induced Adverse Events | From date of radiotherapy started, every 3-4 months within the first 2 years, every 6 months between years 3 and 5, and annually thereafter, assessed up to 100 months.
  Treatment-induced toxicities were scored using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, for events observed after the first dose of irradiation. Toxicities occurred 90 or more days after the completion of CIRT were defined as late toxicities.

SECONDARY OUTCOMES:
Local-progression free survival rate | From date of radiotherapy started until the date of first documented local disease progression, assessed up to 100 months.
  Local-progression free survival rate was defined from the start of carbon ion radiotherapy till the date of local progression or the last follow-up.
Overall survival rate | From date of radiotherapy started until the date of death from any cause, assessed up to 100 months.
  Overall survival rate was defined from the start of carbon ion radiotherapy till the date of death or the last follow-up.
Cause-specific survival rate | From date of radiotherapy started until the date of death caused by thymus tumor treated in this study , assessed up to 100 months.
  Cause-specific survival rate was defined from the start of carbon ion radiotherapy till the date of death caused by thymus tumor treated in this study or the last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jingfang Mao, PHD, Principal Investigator — Shanghai Proton and Heavy Ion Center
Locations (1):
- Shanghai Proton and Heavy Ion Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided